CLINICAL TRIAL: NCT00358709
Title: Treating Psychotic Symptoms of Young Individuals Presenting a First Episode of Schizophrenia: Comparison of Cognitive-Behavioral Therapy and Skills Training Symptom Management on Measures of Symptoms and on Other Indices of Well-Being
Brief Title: Treating Psychotic Symptoms of Young Individuals Presenting a First Episode of Schizophrenia: Comparison of Two State-of-the-Art Interventions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Tania Lecomte, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B02-0769
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
Keywords: Cognitive-behavioral therapy; symptom management; first psychotic episode
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Behavioral Therapy; Palliative Care

INTERVENTIONS:
Behavioral: Cognitive-Behavioral therapy and Symptom Management — A group cognitive-behavioral therapy approach to lessening psychotic symptoms of individuals with a first episode of psychosis, and comparison its effects to a known skills training approach and a control group.

SUMMARY:
To verify the efficacy of a group cognitive-behavioral therapy approach to lessening psychotic symptoms of individuals with a first episode of psychosis, and to compare its effects to a known skills training approach and a control group. Our primary hypotheses were that CBT would do better than the control group at all points in time, and better than the skills training approach, though only at follow-ups

DETAILED DESCRIPTION:
The study's protocol has the following objectives: to verify the efficacy of a group CBT approach; to compare the effects of CBT to those of the symptom management module and to a control group on psychotic symptoms and subjective experiences (e.g., depression, anxiety, self-esteem, social support, insight, and coping); and to assess what the effects are related to, via measuring client variables, therapist variables, and intervention variables that might explain the results. This study follows a randomized controlled trial design where participants are randomly assigned to one of the three groups at each recruiting wave. Both treatment modalities hold the same number of group meetings as well as similar formats, lengths of treatment and operational structures, each operationalized in detailed manuals. Interviewers are blind to group allocation. Symptoms, both psychotic and otherwise, depression, self-esteem, social adaptation, anxiety, insight, social support, and coping are all measured before the beginning of treatment, three months follow-up, nine-months follow-up, and 15-months follow-up

ELIGIBILITY:
Inclusion Criteria:

1) less than two years since their first consultation in psychiatry for psychotic symptoms, 2) a DSM-IV diagnosis in the schizophrenia spectrum (or a psychotic episode suggesting a non-mood related psychosis), 3) ability to read and write in English, 4) aged between 18 and 35, 5) no organic disorder, and 6) consenting to participate

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Estimated)
Dates: Start 2002-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Expected effects on symptoms, measured before beginning of treatment, three months, nine-months, and 15-months follow-ups | 15 months

SECONDARY OUTCOMES:
Self-esteem, social adaptation, coping, insight, substance abuse, measured before beginning treatment, three months, nine-months, and 15-months follow-ups | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Tania Lecomte, Principal Investigator — The University of British Columbia
Locations (1):
- Fraser Health Authority, Surrey, British Columbia, Canada